CLINICAL TRIAL: NCT00005707
Title: Improving Hypertension Care for Inner City Minorities
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4916; R01HL051121 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To improve long-term blood pressure BP) control in a predominantly African-American, low SES community of a large city.

DETAILED DESCRIPTION:
BACKGROUND:

The study was in response to a demonstration and education initiative, "Improving Hypertensive Care for Inner City Minorities", which was reviewed and approved by the Clinical Applications and Prevention Advisory Committee in April 1992 and by the National Heart, Lung, and Blood Advisory Council in May 1992. The Request for Applications was released in October 1992.

DESIGN NARRATIVE:

Components of the program included a community education campaign, an educational intervention for private physicians, and major modifications in the process of care for hypertensives in a health care system that was the largest single provider to the target area. The intervention area was compared to a similar community in another part of the city which was served by different private and public providers. Pre- and post-intervention random samples of persons ages 18-74 were selected from each geographical area to assess the effectiveness of the program in reducing the prevalence of uncontrolled hypertension. The community intervention focused on improving awareness and need to maintain treatment. The private physician intervention focused on strategies for promoting long-term patient adherence. The public hospital clinic/systems components were: 1) educating providers, 2) instituting an evening clinic for the working poor, 3) providing tailored patient education programs which were culturally sensitive and did not require class attendance, and 4) implementing a program in the public hospital emergency center to identify and refer patients with undetected hypertension or hypertension not under regular care.

Efforts, including reminders and follow-up by community health center social workers, were used to keep patients active in treatment programs. The community intervention was directed by the co-investigator from Texas Southern University (TSU), an historically Black university located in the intervention area. He had extensive experience in community outreach. The intervention toward private physicians was directed by investigators from Baylor College of Medicine who had established clinical credibility in the physician community. The investigators from Baylor also had direct supervision over the physicians who provided care in the Harris County Hospital District (HCHD) public health care system. The HCHD was deeply committed to the project and had a high level of representation in all the planning phases.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1998-08

REFERENCES:
- [Background] Hyman DJ, Pavlik VN, Vallbona C, Dunn JK, Louis K, Dewey CM, Wieck L. Blood pressure measurement and antihypertensive treatment in a low-income African-American population. Am J Public Health. 1998 Feb;88(2):292-4. doi: 10.2105/ajph.88.2.292. PMID 9491026
- [Background] Wieck KL. Hypertension in an inner-city minority population. J Cardiovasc Nurs. 1997 Jul;11(4):41-9. doi: 10.1097/00005082-199707000-00005. PMID 9200018